CLINICAL TRIAL: NCT01492075
Title: Phase IV Study of Postoperative Pain Management
Brief Title: A Comparison Between Continuous and Intermittent Intraabdominal Analgesia Using Local Anaesthetics
Acronym: PoPuLAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Anil Gupta, Associate Professor, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20100101
Record Dates: First submitted 2011-10-07; First posted 2011-12-14 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Abdominal Hysterectomy
Keywords: Postoperative pain; Anesthetics: Local anesthetics; Surgery: Hysterectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous infusion (Active Comparator): Continuous infusion of LA intraabdominally
  Interventions: Drug: PCRA (Intermittent injection)
- PCRA (Intermittent injection) (Experimental): Patient controlled LA intraabdominally
  Interventions: Drug: PCRA (Intermittent injection)

INTERVENTIONS:
Drug: PCRA (Intermittent injection) — Intermittent injection of LA intraabdominally

SUMMARY:
The investigators hypothesis is that patient controlled local anesthetics administered intraabdominally are more efficacious compared to continuous infusion in reducing postoperative pain and morphine consumption.

DETAILED DESCRIPTION:
Open abdominal hysterectomy is a common procedure performed for many benign and malignant gynaecological diseases and is associated with moderate to severe pain. Traditional methods for postoperative pain management include patient controlled intravenous analgesia (PCA) using morphine, epidural analgesia and spinal analgesia with opiates but recently, even local aesthetic (LA) has been used intra-abdominally and into the abdominal wall. Although epidural analgesia may be considered by some to be gold standard for pain relief following abdominal surgery, a recent publication and past experience over several years may question the use of invasive techniques for lower abdominal surgery. Thus, there is a trend towards movement from central blocks towards other non-invasive methods for pain relief.

PCA with morphine is now commonly used for management of pain following major surgery and compared to central blocks, has advantages in being relatively safe, easy to use and associated with a high degree of patient satisfaction. However, the large doses of morphine necessary to ensure adequate postoperative analgesia means that side effects such as postoperative nausea and vomiting (PONV), tiredness, pruritus, headache and constipation may be a major problem in this group of patients. Therefore, alternative techniques to reduce morphine requirements are increasingly being used. These include the use of paracetamol, non-steroidal anti-inflammatory drugs (NSAID) and recently local anaesthetics (LA). The latter have been found to result in morphine sparing by 30 - 40 % and even a reduction in postoperative nausea (PON). LA infused intraperitoneally is safe and effective and a recent study showed that using 12.5 mg/h levobupivacaine could attain adequate analgesia. Thus, efficacy of LA has been established as well as the dose. However, the method of administration of LA intraperitoneally remains unclear.

This study is designed with the primary aim of studying whether morphine consumption can be reduced postoperatively using the patient-controlled administration system for intraperitoneal LA compared to a continuous infusion, and whether this translates into improved recovery parameters or reduced side effects and improved patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. 18 -65 year old patients undergoing open abdominal hysterectomy.
2. ASA I - II (Appendix 1).
3. Have signed and dated Informed Consent.
4. Willing and able to comply with the protocol for the duration of the trial.

Exclusion Criteria:

1. Patients undergoing open abdominal hysterectomy due to suspected cancer.
2. Patients with chronic pain who are taking analgesics regularly.
3. Allergy to components in levobupivacaine (Chirocaine)/Saline (Sodium Chloride).
4. Participation in other clinical trials.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 0-24 h
  Total morphine consumption 0 - 24 h postoperatively

SECONDARY OUTCOMES:
Postoperative pain | 0 - 48 h postoperatively
  Post-operative pain assessed on the basis of NRS (Numeric Rating Score).
PONV | 0 - 48 h postoperatively
  Incidence of nausea and vomiting and anti-emetic requirement
Home discharge | 0-10 days
  Time to home readiness and time to return to work.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Perniola, MD, Principal Investigator — Örebro University, Sweden; Anil Gupta, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- University Hospital, Örebro, Sweden